CLINICAL TRIAL: NCT03653780
Title: Physiological Responses During Overground Gait Training With a Wearable Exoskeleton After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Nina Lefeber, Doctoral Researcher, Vrije Universiteit Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EKSO STUDY II
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Stroke
Keywords: Wearable Exoskeleton; Stroke; Oxygen Consumption; Cardiorespiratory Responses
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ekso GT gait training (Experimental): 20-minute Ekso GT gait training
  Interventions: Device: Ekso GT

INTERVENTIONS:
Device: Ekso GT — Walking in the Ekso GT with maximum bilateral assistance for 20 minutes

SUMMARY:
To investigate the acute physiological responses during 20-minute overground gait training with a wearable exoskeleton in persons after stroke

DETAILED DESCRIPTION:
STUDY DESIGN: An experimental, 1-group trial

PATIENT RECRUITMENT: A minimum of 10 subjects will be included in the study. Patients will be recruited at the Revarte Rehabilitation Hospital (Edegem, Belgium).

ELIGIBILITY CRITERIA: see section "Eligibility"

PROCEDURES: The trial will be conducted at the Revarte Rehabilitation Hospital (Edegem, Belgium).

Before the start of the study, informed consent and baseline patient characteristics will be collected.

On a separate day before the start of the 5th training session, patients will be seated for 5 minutes during which resting values (respiratory gases and heart rate) will be assessed.

Next, participants will be measured during their 5th training session with the Ekso GT with maximum bilateral assistance. Following settings will be used: sitting program ("Min lean"); standing program ("Auto lean"); step initiation program ("ProStep+"), training mode ("Both"), assistance mode ("Bilat"), swing assistance ("Max"), stance support ("Full").

At the start of the 5th training, a mouth mask, heart rate monitor and gait analysis system will be applied. After a seated resting period of 5 minutes, patients will walk for a total of 20 minutes during which respiratory gases and heart rate will be monitored continuously. The Borg rating of perceived exertion will be registered every 5 minutes. The intervention will be terminated early when relative or absolute indications are presented as reported by the American Heart Association or when patients are unable to continue walking.

During training, patients will walk at a self-selected walking speed.

RESTRICTIONS & PROHIBITIONS: Participants will be instructed to not consume food, alcohol, caffeine or nicotine at least 3h prior to the intervention. Usual medication intake will be allowed with small amounts of water.

MATERIALS: During the overground gait training sessions, the Ekso GT robotic exoskeleton with SmartAssist (Ekso Bionics Inc., USA) will be used. A flexible facemask (adult facemask, small/medium, Cortex, Germany), lightweight chest carrying gas analysis system (Metamax 3B, Cortex, Germany) and Bluetooth heart rate belt (Polar H7, Polar Electro, Finland) will be used to measure metabolic and cardiorespiratory parameters. At the start of each measurement, gas (room air and reference gas (17.4% O2 and 5.1% CO2)) and volume (3L syringe) calibrations of the breath-by-breath gas analysis system will be performed in accordance with the manufacturer's instructions.

OUTCOMES: See section "Outcome measures"

ELIGIBILITY:
Included will be persons who

* Had a stroke (1 week to 6 months since injury)
* Are 18 years or older
* Cannot walk independently or can walk independently on level ground, but require help on stairs, slopes or uneven surfaces (FAC 0 - 4)
* Have prior experience with the Ekso GT (i.e. 4 training sessions)

Excluded will be persons who

* Can walk independently on level ground, stairs, slopes and uneven surfaces (FAC = 5)
* Have musculoskeletal problems (other than stroke) affecting the ability to walk
* Have concurrent pulmonary diseases (e.g. asthma)
* Have unstable cardiovascular conditions
* Have concurrent neurological diseases (e.g. Parkinson's Disease)
* Have communicative and/or cognitive problems affecting the ability to understand or follow instructions
* Present contra-indications for using the Ekso GT (according to manufacturer's instructions)

  * Severe concurrent medical diseases (infections, circulatory, heart or lung, pressure sores)
  * Severe spasticity (Ashworth 4)
  * Range of motion restrictions that would prevent a patient from achieving normal, reciprocal gait pattern, or would restrict a patient from completing normal sit-to-stand or stand-to-sit transitions

    * Bilateral hip flexion < 110°
    * Knee flexion contracture > 12°
    * Inability to achieve 0° neutral angle dorsiflexion with knee flexion ≤ 12°
  * Weight ≥ 100 kg
  * Hip width < 35.8 cm or > 45.6 cm
  * Upper leg length < 51 cm or > 61.4 cm
  * Lower leg length < 48 cm or > 63.4 cm
  * Upper leg length discrepancy > 0.5 inch (1.3 cm)
  * Lower leg length discrepancy > 0.75 inch (1.9 cm)
  * Unstable spine, unhealed limbs or pelvic fractures
  * Unhealthy bone density
  * Heterotopic ossification
  * Significant contractures
  * Elbows and shoulders cannot support crutches, walker or cane
  * Psychiatric or cognitive situations that may interfere with proper operation of the device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Net oxygen cost (OC, ml/kg/m) at minute 5 of walking | Minute 5 of 20-minute walking period
  Net oxygen consumption (oxygen consumption (ml/kg/min) during walking minus during rest) divided by the walking speed (m/min)
Net oxygen cost (OC, ml/kg/m) at minute 10 of walking | Minute 10 of 20-minute walking period
  Net oxygen consumption (oxygen consumption (ml/kg/min) during walking minus during rest) divided by the walking speed (m/min)
Net oxygen cost (OC, ml/kg/m) at minute 15 of walking | Minute 15 of 20-minute walking period
  Net oxygen consumption (oxygen consumption (ml/kg/min) during walking minus during rest) divided by the walking speed (m/min)
Net oxygen cost (OC, ml/kg/m) at minute 20 of walking | Minute 20 of 20-minute walking period
  Net oxygen consumption (oxygen consumption (ml/kg/min) during walking minus during rest) divided by the walking speed (m/min)
Net heart rate (HR, beats/min) at minute 5 of walking | Minute 5 of 20-minute walking period
  Heart rate during walking (beats/min) minus resting heart rate
Net heart rate (HR, beats/min) at minute 10 of walking | Minute 10 of 20-minute walking period
  Heart rate during walking (beats/min) minus resting heart rate
Net heart rate (HR, beats/min) at minute 15 of walking | Minute 15 of 20-minute walking period
  Heart rate during walking (beats/min) minus resting heart rate
Net heart rate (HR, beats/min) at minute 20 of walking | Minute 20 of 20-minute walking period
  Heart rate during walking (beats/min) minus resting heart rate
Net minute ventilation (VE, L/min) at minute 5 of walking | Minute 5 of 20-minute walking period
  The amount of air in- or exhaled per minute (L/min) during walking minus during rest
Net minute ventilation (VE, L/min) at minute 10 of walking | Minute 10 of 20-minute walking period
  The amount of air in- or exhaled per minute (L/min) during walking minus during rest
Net minute ventilation (VE, L/min) at minute 15 of walking | Minute 15 of 20-minute walking period
  The amount of air in- or exhaled per minute (L/min) during walking minus during rest
Net minute ventilation (VE, L/min) at minute 20 of walking | Minute 20 of 20-minute walking period
  The amount of air in- or exhaled per minute (L/min) during walking minus during rest
Net respiratory exchange ratio (RER, no unit) at minute 5 of walking | Minute 5 of 20-minute walking period
  The ratio between the amount of CO2 produced by the body and the amount of VO2 consumed by the body minus the ratio at rest
Net respiratory exchange ratio (RER, no unit) at minute 10 of walking | Minute 10 of 20-minute walking period
  The ratio between the amount of CO2 produced by the body and the amount of VO2 consumed by the body minus the ratio at rest
Net respiratory exchange ratio (RER, no unit) at minute 15 of walking | Minute 15 of 20-minute walking period
  The ratio between the amount of CO2 produced by the body and the amount of VO2 consumed by the body minus the ratio at rest
Net respiratory exchange ratio (RER, no unit) at minute 15 of walking | Minute 20 of 20-minute walking period
  The ratio between the amount of CO2 produced by the body and the amount of VO2 consumed by the body minus the ratio at rest

SECONDARY OUTCOMES:
Net Rating of Perceived Exertion (RPE, 6-20) at minute 5 of walking | Minute 5 of 20-minute walking period
  Rating of perceived effort, strain and/or fatigue during walking, pointed on a 15-point Borg scale (6-20) during walking minus during rest
Net Rating of Perceived Exertion (RPE, 6-20) at minute 10 of walking | Minute 10 of 20-minute walking period
  Rating of perceived effort, strain and/or fatigue during walking, pointed on a 15-point Borg scale (6-20) during walking minus during rest
Net Rating of Perceived Exertion (RPE, 6-20) at minute 20 of walking | Minute 15 of 20-minute walking period
  Rating of perceived effort, strain and/or fatigue during walking, pointed on a 15-point Borg scale (6-20) during walking minus during rest
Net Rating of Perceived Exertion (RPE, 6-20) at minute 20 of walking | Minute 20 of 20-minute walking period
  Rating of perceived effort, strain and/or fatigue during walking, pointed on a 15-point Borg scale (6-20) during walking minus during rest

OTHER OUTCOMES:
Walking speed (m/min) at minute 5 of walking | Minute 5 of 20-minute walking period
  The distance (meters) walked per minute
Walking speed (m/min) at minute 10 of walking | Minute 10 of 20-minute walking period
  The distance (meters) walked per minute
Walking speed (m/min) at minute 15 of walking | Minute 15 of 20-minute walking period
  The distance (meters) walked per minute
Walking speed (m/min) at minute 20 of walking | Minute 20 of 20-minute walking period
  The distance (meters) walked per minute

CONTACTS AND LOCATIONS:
Overall Officials: Eric Kerckhofs, PhD, Study Chair — Vrije Universiteit Brussel; Eva Swinnen, PhD, Study Director — Vrije Universiteit Brussel; Nina Lefeber, PhD student, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- RevArte Rehabilitation Hospital, Edegem, Antwerp, Belgium